CLINICAL TRIAL: NCT06999161
Title: Therapeutic Drug Monitoring of Beta-lactams and Renal Hyperclearance in Patients Admitted to Intensive Care for Acute Brain Injury
Acronym: BETALACT-ARC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2025/CR-01
Record Dates: First submitted 2025-05-13; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Brain Injuries
Keywords: Beta-Lactams; Renal Clearance; Therapeutic Drug Monitoring
MeSH Terms: conditions — Critical Illness; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BETALACTAM Treated Patients: Adult patients (≥18 years) admitted to intensive care for acute brain injury, presenting with an infectious episode, documented augmented renal clearance (as assessed by urinary creatinine clearance), and receiving treatment with beta-lactam antibiotics.

SUMMARY:
Augmented Renal Clearance (ARC), defined as a supraphysiological increase in renal function, is frequently observed in critically ill patients, particularly those with acute brain injury. ARC complicates the management of renally eliminated drugs, specifically beta-lactam antibiotics, by enhancing drug clearance and thereby increasing the risk of underdosing and therapeutic failure. Although pharmacological therapeutic drug monitoring (TDM) is recommended to optimize dosing, it remains limited by issues of accessibility, highlighting the need for alternative approaches to identify at-risk patients and adjust dosing based on renal function.

Early identification of patients at risk for subtherapeutic beta-lactam plasma concentrations could enable timely dose adjustments. A combined assessment of renal function and beta-lactam TDM could enhance our understanding of the kinetics of both parameters. These data may support the development of predictive models capable of proposing individualized dosing regimens based on renal function.

Optimizing beta-lactam plasma concentrations in this patient population could improve infection management and potentially enhance clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Admitted to the intensive care unit for acute brain injury
* Exhibiting Augmented Renal Clearance (ARC), defined by a urinary creatinine clearance (ClCrU) greater than 130 mL/min/1.73 m² on at least one measurement
* Receiving Therapeutic Drug Monitoring (TDM)-guided treatment with one of the following beta-lactam antibiotics: amoxicillin/clavulanic acid, cefotaxime, piperacillin/tazobactam, cefepime, or meropenem
* Affiliated with or benefiting from a health insurance scheme

Exclusion Criteria:

* Estimated life expectancy <24 hours
* Patients who have expressed opposition to study participation
* Patients under legal protection (guardianship, curatorship, or court protection)
* Patients currently in an exclusion period determined by participation in another study
* Patients already enrolled in a study that precludes concurrent participation in an observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied included patients admitted to the intensive care unit with acute brain injury (of traumatic, vascular, infectious or immunological origin), presenting a profile of HCR and receiving antibiotic treatment with betalactam
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma betalactam underdosing | 24 hours after the start of antibiotic therapy, and repeated every 48 hours or in the event of underdosing, overdosing, change of molecule or significant variation in renal function, assessed until the antibiotic therapy is stopped, for up to 14 days
  Development of a predictive model for plasma beta-lactam underdosing in critically ill patients with acute brain injury and renal hyperclearance, receiving beta-lactam therapy for an ongoing infectious episode.
  Plasma beta-lactam concentrations will be measured 24 hours after initiation of antibiotic therapy, and subsequently every 48 hours, or in cases of underdosing, overdosing, antibiotic switch, or significant changes in renal function.

SECONDARY OUTCOMES:
Evolution of Augmented Renal Clearance | From date of inclusion until the date of discharge from intensive care, assessed up to 28 days
  Assessment of urinary creatinine clearance based on urine collection (8, 12, or 24-hour collection depending on center practices).
Evolution of plasma Beta-lactam Concentration | From date of inclusion until the date of discharge from intensive care, assessed up to 28 days
  Monitoring of total plasma beta-lactam concentrations obtained through Therapeutic Drug Monitoring during the intensive care stay
Relationship Between Plasma Underdosing Intensity and Level of Augmented Renal Clearance (ARC) | From date of inclusion until the date of discharge from intensive care, assessed up to 28 days
  Characterization of the intensity of plasma beta-lactam underdosing for each antibiotic molecule relative to the degree of ARC.
Beta-lactam Dosing According to Augmented Renal Clearance Level. | From date of inclusion until the date of discharge from intensive care, assessed up to 28 days
  Development of a dosing nomogram for beta-lactam antibiotics tailored to the degree of ARC.
Clinical outcome | From date of inclusion until the date of discharge from intensive care, assessed up to 28 days
  Assessment of clinical outcomes based on rates of clinical success and failure.
  * Clinical success is defined as the resolution of infectious symptoms present at the initiation of antibiotic therapy, allowing discontinuation of antibiotics at the end of the planned treatment duration.
  * Clinical failure is defined as the persistence or worsening of initial symptoms, the occurrence of superinfection (infection with newly identified pathogens), or recurrence (a new infectious episode with the same pathogen).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided